CLINICAL TRIAL: NCT02308774
Title: Osteomyelitis: Procalcitonin to Diagnose and Monitor Osteomyelitis
Brief Title: Osteomyelitis: Procalcitonin to Diagnose and Monitor Osteomyelitis (PCT)
Acronym: PCT
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 022014-007
Record Dates: First submitted 2014-11-07; First posted 2014-12-04 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Osteomyelitis
Keywords: osteomyelitis, diabetic foot infection
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
We plan a cohort study of 40 diabetic patients admitted to Parkland hospital with a foot infection. We will enroll a representative cross section of subjects with diabetic foot infection. Patient will be consented and will receive therapy based on standard protocols. Currently patients with suspected osteomyelitis have bone biopsies to identify bacterial pathogens and verify MRI diagnosis. Repeat bone biopsies are performed at the end of therapy to verify that osteomyelitis has been successfully treated. Serum to measure procalcitonin will be obtained at baseline, week 3 and week 6.

DETAILED DESCRIPTION:
Infection: will be defined as a patient with three of six clinical signs of infection (erythema, heat, edema, pain, loss of function, purulence) or leukocytosis. We will use the Infectious Diseases Society of America's Diabetic Foot Infection guidelines to stratify the severity of infection. This guideline stratifies infections into three categories (mild, moderate, and severe) based on practical clinical and laboratory findings. Our group has shown this system to be predictive of morbidity.

Osteomyelitis Diagnosis: We will evaluate suspected cases of osteomyelitis with bone biopsy for histology and culture and sensitivity. Bone biopsy to diagnose osteomyelitis is part of the standards of care established from the "diabetic foot infection guidelines" in our institution. We expect 1/4 of patients will have negative bone biopsy results. We will define a positive case of osteomyelitis as bone with positive bacterial cultures or histologic finding of acute osteomyelitis or chronic osteomyelitis. Acute osteomyelitis will be defined as the presence of acute inflammatory cells, congestion or thrombosis of medullary or periosteal small vessels, and necrotic bone. Chronic osteomyelitis will demonstrate areas of woven bone and fibrosis with large numbers of lymphocytes, histiocytes, and plasma cells.

Outcome Measures: Our primary endpoints will be resolution of osteomyelitis based on percutaneous bone biopsy six weeks after initiation of therapy. We will evaluate patients for six months for signs of recurrent osteomyelitis and other clinical outcomes (wounds, Charcot fracture, and infection). Clinical outcomes will include (1.) wound healing, (2.) limb salvage, (3.) hospitalizations for recurrent diabetic foot infection (4.) surgical procedures, and (5.) recurrent ulcers.

Confounding Variables: Most imaging studies of diabetic foot osteomyelitis do not assess potential confounding variables such as wound severity, diabetes severity, diabetes co-morbidities, and perfusion to the extremity. Outcomes such as wound healing and resolution of infection are clearly affected by current medical problems, social history, peripheral arterial disease, wound severity, and treatment factors such as type of antibiotics, off-loading, debridement and vascular surgery interventions. We will include the following variables in the study and in the analysis plan.

1. Medical History: The diagnosis of diabetes will be based on American Diabetes Association criteria. We will evaluate glycated hemoglobin at baseline and quarterly per our standard of care. In addition, we will document: duration and type of diabetes, type of diabetes medication (insulin, oral, combination therapy, diet), previous history of foot ulcers, amputation (toe, foot), lower extremity bypass, lower extremity angioplasty, Coronary artery bypass surgery, cardiac angioplasty, arthritis, liver disease, osteoporosis, malignancy, and bone tumors. We will use the Kaplan co-morbidity index to record disease severity. We will use the New York Heart Association criteria to classify congestive heart failure, and the National Kidney Foundation Disease Outcomes Quality Initiative Clinical Practice Guidelines for chronic kidney disease to stage kidney disease. We will measure height and weight to determine body mass index (BMI). We will document all prescription and over-the-counter medications as well as the type, route and duration of antibiotic therapy.
2. Social Factors: We will evaluate the following factors: marital status, years of education, type of work, tobacco history (pack years, current smoker, current use of chewing tobacco, previous smoker, no tobacco history), drug history (current, previous history, no drug history), and alcohol history.
3. Vascular Assessment: We will assess perfusion of the macro-circulation with arterial Doppler studies and micro-circulation with Skin Perfusion Pressure measurements.
4. Wound Assessment: We will use the University of Texas Diabetic Ulcer Classification to grade ulcer severity. We use acetate tracings, clinical measurements of length, width and depth and digital photos to measure wound area and volume before and after debridement. These technique has been shown to be highly reproducible. A wound will be considered "healed" when it is fully epithelialized with no drainage.
5. Offloading and Debridement: For wounds on the weight-bearing surface of the foot, the most feasible offloading modality will be provided based on postural stability, wound location, and patient acceptance. Modalities available will be total contact cast, removable boot, healing sandal, and therapeutic shoes. Debridement will be performed as needed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Age ≥ 21 years
* Infectious Disease Society of America stage 3 infection

Exclusion Criteria:

* History of previous bone infection in the study foot
* Unable to provide informed consent
* HIV, Hepatitis, osteomyelitis at other sites

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified from the investigator's inpatient and outpatient populations. This is not a treatment study, so subjects participating in other protocols will also be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoints will be changes in procalcitonin levels at Baseline, Week 3 and Week 6 correlated with resolution of osteomyelitis based on percutaneous bone biopsy six weeks after initiation of therapy. | 6 weeks
  Serial measurements of procalcitonin at Baseline, Week 3 and Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States